# **Evaluation of the Efficacy of Different Drugs in the Treatment of Pain in Patients with Temporomandibular Disorder**

Levent Ciğerim DDS, PhD 1, Mehmet Güzel1, Zeynep Dilan Orhan1

<sup>1</sup> Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial

Surgery, Van, TURKEY

Corresponding author: Levent Ciğerim

Address: Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial

Surgery, Van, Turkey Postal Code: 65080

E-mail address: levent139@hotmail.com Phone:+905321633287 Office Phone: 904322251744

Fax: +904322251747

#### Levent CİĞERİM

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery levent139@hotmailmail.com, +905321633287, https://orcid.org/0000-0001-5218-8568

## Mehmet GÜZEL

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:dtmehmetguzel@gmail.com">dtmehmetguzel@gmail.com</a>, +905363609854, <a href="https://orcid.org/0000-0002-9621-0496">https://orcid.org/0000-0002-9621-0496</a>

#### Zeynep Dilan Orhan

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:zeynepdilanorhan@gmail.com">zeynepdilanorhan@gmail.com</a>, +905425525525, <a href="https://orcid.org/0000-0003-1333-9073">https://orcid.org/0000-0003-1333-9073</a>

#### **Study Protocol, Methods and Procedures to be Applied:**

The study is planned to be carried out on 200 patients aged 18 and over, who applied to Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, with complaints of pain due to tempromandibular disease. When patients first apply to the clinic, their anamnesis will be taken and they will be directed to mr imaging after clinical evaluation. Patients who meet the inclusion criteria and volunteer will be included in the study. Patients will be randomly divided into 4 groups. Medications will be given to patients by auxiliary staff and the study will be double-blind.

Medicines will be given as follows. Dexketoprofen Trometamol + Thiocolchicoside (25mg + 4mg, 2x1) in the 1st group, Dexketoprofen Trometamol + Paracetamol (25mg + 300mg, 2x1) in the 2nd group, only Dexketoprofen Trometamol (25mg, 2x1) in the 3rd group and paracetamol 500 in the 4th control group. mg (4x1) will be given. In addition, patients in each group will use the occlusal plate with study drugs for a maximum of 8 hours per day (at night). Medicines will be used regularly for 2 weeks. Paracetamol 500 mg will be used with the occlusal plate for the next 2 weeks, only if needed. The pain values of the patients will be evaluated with the VAS scale, and the amount of mouth opening will be evaluated by measuring the distance between the incisal edges of the lower and upper central teeth. Follow-up and controls of the patients will be done in the preoperative period, at the 2nd and 4th weeks postoperatively, and the findings will be recorded. After the 1st month, the patients will be followed up to the 3rd month and the treatment of those who need additional treatment will be continued.

Obtained data will be analyzed and evaluated statistically.

### **Statistical Data Analysis:**

Deviation, Minimum and Maximum values; will be expressed as numbers and percentages for categorical variables. Mann-Whitney U analysis will be used to compare group means in terms of continuous independent variables. In addition, the Wicoxon test will be calculated in the comparison of double dependent groups. In order to determine the relationship between these variables, Spearman correlation coefficients will be calculated separately for the groups. Chi-square test will be used to determine the relationship between groups and categorical variables. Statistical significance level will be taken as 5% in calculations and SPSS statistical package program will be used for calculations.